CLINICAL TRIAL: NCT07231679
Title: A Randomized, Placebo-Controlled, Multicenter, Phase 1/2a Study to Investigate the Safety, Tolerability, and Pharmacokinetics of IGT-303 in Healthy Volunteers and Participants With Chronic Kidney Disease
Brief Title: A Study to Investigate IGT-303 in Healthy Volunteers and Participants With Chronic Kidney Disease
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ingenia Therapeutics INC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IGT-303-01-CKD01
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteers; Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IGT-303 (Experimental): Part A: single ascending dose (SAD), 6 cohorts Part B: multiple ascending dose (MAD), 3 cohorts
  Interventions: Drug: IGT-303
- Placebo (Placebo Comparator): Placebo (normal saline)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IGT-303 — IGT-303 administered via IV or SC
  Arms: IGT-303
Drug: Placebo — Saline
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to observe the safety of IGT-303 in healthy volunteers and participants with Chronic Kidney Disease. The main question it aims to answer is:

Is IGT-303 safe as a single dose or multiple dose regimen when applied under the skin (subcutaneously (SC)) or to a vein (intravenously (IV)).

Researchers will compare IGT-303 against a placebo to see if IGT-303 is safe for use.

Participants will be assigned to either IGT-303 or placebo and assessed for safety and tolerability for the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant 18-60 years of age, inclusive, at Screening;
* Able to understand the key components of the study as described in the written informed consent document, and willing and able to provide written informed consent;
* Body mass index (BMI) within the range of 18.5 to 32 kg/m2 at Screening;
* Participants assigned male at birth (AMAB) will be either sterile or agree to use an approved method of contraception from Screening until at least 5 half-lives plus 90 days after the last dose of study drug, or do not engage in sexual relations which carry a risk of pregnancy (does include abstinence), and agree to refrain from sperm donation and in vitro fertilization until 5 half-lives plus 90 days after the last dose of the study drug;
* In the opinion of the Investigator, is able to adhere to the requirements of the study, including required overnight stays in the research site.

Exclusion Criteria:

* Known allergy to study medication or its components (non-medicinal ingredients) or a history of a severe allergic reaction to any drug or history of multiple food/drug allergies;
* Use of cigarettes exceeding >5 cigarettes per week at time of Screening; social/casual cigarette use (≤5 per week) is permitted during the study, but participants must be willing to abstain during inpatient confinement;
* Positive urine screen for drugs of abuse including tetrahydrocannabinol or has a positive breathalyzer test, at Screening or at Day -1;
* Any illness or medical history that would impact safety or compliance with study requirements or impact ability to interpret study data.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Estimated)
Dates: Start 2025-10-30 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs), serious adverse events (SAEs), and treatment-emergent adverse events (TEAEs) | From Screening to Day 84.
  The number and severity (by Grade) will be measured.

SECONDARY OUTCOMES:
PK Parameters of Intravenous (IV) and Subcutaneous (SC) IGT-303 | Day 1 to Day 84.
  Maximum observed concentration (Cmax)
PK Parameters of IV and SC IGT-303 | Day 1 to Day 84
  Observed time of maximum concentration (Tmax)
PK Parameters of IV and SC IGT-303 | Day 1 to Day 84
  Terminal exponential rate constant, determined using the linear least squares regression of the terminal phase of the log-serum concentration time profile (λz)
PK Parameters of IV and SC IGT-303 | Day 1 to Day 84
  Terminal exponential half-life, calculated as ln(2)/λz (T1/2)
PK parameters of IV and SC IGT-303 | Day 1 to Day 84
  Area under the concentration-time curve calculated using linear trapezoidal rule from time zero to time t, where t is the time of the last observed quantifiable concentration (AUC0-t)
PK parameters of IV and SC IGT-303 | Day 1 to Day 84
  Area under the concentration-time curve from time zero to infinity, defined as AUC0-t + Ct/λz (AUC0-∞)
PK parameters of IV and SC IGT-303 | Day 1 to Day 84
  Total clearance (CL), defined as dose/AUC0-∞
PK parameters of IV and SC IGT-303 | Day 1 to Day 84
  Terminal volume of distribution (Vz), defined as CL/λz
PK parameters of IV and SC IGT-303 | Day 1 to Day 84
  Absolute bioavailability (F), defined as the dose-corrected (AUC0-∞ SC) / (AUC0-∞ IV)

CONTACTS AND LOCATIONS:
Overall Officials: Emma Trowbridge, MD, Principal Investigator — Nucleus Network
Locations (1):
- Nucleus Network, Herston, Brisbane, Australia

IPD SHARING:
Plan to Share IPD: No